CLINICAL TRIAL: NCT07048067
Title: Ultrasound Evaluation for Baxter VASCU-GUARD Vascular Patches Post-Endarterectomy and Complications Assessment
Acronym: VASCU-GUARD
Status: Completed | Type: Observational
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Rahimi, Maham, Associate Professor of Cardiovascular Surgery, The Methodist Hospital Research Institute
Other Study IDs: 00038233
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Carotid Endarterectomy (CEA) Surgical Patients
Keywords: carotid endarterectomy (CEA); VASCU-GUARD
MeSH Terms: interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients undergoing carotid endarterectomy with the use of VASCU-GUARD vascular patches: Follow-up ultrasound assessment available
  Interventions: Procedure: Carotid endarterectomy (CEA)

INTERVENTIONS:
Procedure: Carotid endarterectomy (CEA) — carotid endarterectomy (CEA) with the use of Baxter VASCU-GUARD vascular patches

SUMMARY:
VASCU-GUARD vascular patches with the new packaging have been available at the Houston Methodist Hospital since January 2023. This study is a retrospective chart review, aiming to compare the performance of Baxter VASCU-GUARD vascular patches implemented during carotid endarterectomies (CEA) prior to January 2023 and after January 2023. This study is one of a kind, as no other comparative retrospective chart review on the performance of VASCU-GUARD vascular patches from the old and new packaging has been published yet.

The project will contribute to the scientific knowledge about long-term outcomes associated with the use of patch material during endarterectomies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above.
* Patients undergoing carotid endarterectomy with the use of VASCU-GUARD vascular patches.
* Follow-up ultrasound assessment available

Exclusion Criteria:

• No postoperative ultrasound assessment is available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing carotid endarterectomy (CEA) with the use of Baxter VASCU-GUARD vascular patches in all campuses of the Houston Methodist Hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Ultrasound evaluation of Baxter VASCU-GUARD vascular patches | 1/1/2023 - 4/30/2024
  Retrospective review of ultrasound recordings and ultrasound reports at one-month, 3-months, 6-months and 1-year follow-up after endarterectomy - if available, to evaluate patch patency, morphology, integrity, complications, and blood flow dynamics

SECONDARY OUTCOMES:
Complications assessment | 1/1/2023 - 4/30/2024
  Analyze complications linked with Baxter Vascular Patches (VASCU-GUARD), including but not limited to thrombosis, stroke, dissection, restenosis, infection, fluid collection, pseudoaneurysm formation, fraying or irregularities in patch material.
Correlation with Clinical Outcomes | 1/1/2023 - 4/30/2024
  Recognize correlations between ultrasound findings and clinical outcomes. This correlation will complement the understanding of how ultrasound monitoring can predict and influence patient prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Only study findings to be shared

DOCUMENTS (1):
  • Study Protocol (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT07048067/Prot_000.pdf